CLINICAL TRIAL: NCT00061230
Title: Efficacy of Relaxation Training
Brief Title: Relaxation Training to Decrease Pain and Improve Function in Adolescents With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P01HD33988-00606A1; P01HD033988 (NIH)
Record Dates: First submitted 2003-05-22; First posted 2003-05-23 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-04

CONDITIONS: Cerebral Palsy
Keywords: Relaxation training
MeSH Terms: conditions — Cerebral Palsy

INTERVENTIONS:
Behavioral: biofeedback-monitored relaxation training

SUMMARY:
This study will examine the effectiveness of relaxation training for providing pain relief and improving physical and psychological functioning in youth with physical disabilities due to cerebral palsy.

DETAILED DESCRIPTION:
Chronic pain is a serious problem in many youths with disabilities. There is a growing body of research supporting the efficacy of relaxation training for reducing chronic pain in adults. Given this evidence, there has been a growing interest in determining whether these findings also generalize to youths with chronic pain. This study will address a significant gap in the medical literature by examining the efficacy of relaxation training for providing pain relief and improving function in youths with physical disabilities. The study will evaluate the effects of relaxation training on global physiological arousal, pain-site specific muscle tension, and perceived control over pain. Physiological arousal will be assessed via hand temperature and galvanic skin response. Muscle tension will be assessed via surface EMG biofeedback recordings before, during, and after each treatment session. Self-efficacy concerning pain control will be assessed via a modified Survey of Pain Attitudes and modified Coping Strategies Questionnaire.

Sixty youth (age range 10 to 20 years old) with spastic type cerebral palsy (CP) will be randomly assigned to either the relaxation training group or a distraction control group. Youths in the relaxation training group will be given eight sessions of autogenic relaxation training and will be asked to practice relaxation at home using audio tapes. Youths in the distraction control group will receive eight sessions of distracting story-telling and will be asked to listen to age-appropriate audio tapes of stories at home. Study visits are scheduled weekly for eight weeks. Average pain intensity will be assessed with a numerical rating scale. Secondary outcome measures include psychological functioning and pain interference with personal activities. Medical services utilization will be assessed by asking the parent or guardian about any medications taken by the participant, any illnesses or medical complications, any medical treatments received, and the frequency of health care visits. Participants will be assessed at 1, 3, 6, 9, and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy
* Referred by the study physician
* Chronic cerebral palsy-related pain for at least 3 months prior to study entry. The pain needs to have an average daily occurrence of 3 on a 0 to 10 scale, where 0 is no pain and 10 is extreme pain.
* Primary language is English

Exclusion Criteria

* Acute painful conditions
* Cognitive impairment as determined by a score < 12 on the modified Mini-Mental Status Exam

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60
Dates: Start 2003-03; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Joyce M. Engel, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States